CLINICAL TRIAL: NCT03674775
Title: Dialogue Around Respiratory Illness Treatment for Family Practice (DART -FP)
Brief Title: Reducing Antibiotic Prescribing in Family Practice
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Rita Mangione-Smith, Professor and Chief, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 371934
Record Dates: First submitted 2018-09-06; First posted 2018-09-18 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Acute Respiratory Tract Infection

STUDY DESIGN:
Intervention Model Description: cluster randomized control trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group Providers (Active Comparator): DART QI Program Participation
  Interventions: Other: DART QI Program Participation
- Control Group Providers (No Intervention): Usual Care

INTERVENTIONS:
Other: DART QI Program Participation — Antibiotic prescribing data will be collected at multiple time points both before and after the initiation of the intervention.
  Arms: Intervention Group Providers

SUMMARY:
Antibiotic prescribing for childhood acute respiratory tract infections (ARTIs), including acute otitis media (AOM), pharyngitis, sinusitis, bronchitis, and upper respiratory infection (URI), is common in the United States (US). In the outpatient setting, more than 50% of children diagnosed with ARTIs receive antibiotic prescriptions. Considering that the estimated US prevalence of pediatric bacterial ARTIs is 27% (with the remainder of ARTIs caused by viruses) this represents a substantial degree of antibiotic overuse nationwide. Another troubling trend in antibiotic prescribing for ARTIs in children is the increased reliance on broad-spectrum, second-line agents for bacterial ARTIs. Unwarranted use of antibiotics, especially broad-spectrum agents, has been associated with increased resistance among several strains of bacteria that commonly cause ARTIs, posing risks to both individuals and communities.

DETAILED DESCRIPTION:
Provider-parent communication during ARTI visits often drives unwarranted antibiotic prescribing. Dr. Mangione-Smith (proposed principal investigator) and colleagues developed a quality improvement (QI) intervention for pediatric providers called the Dialogue Around Respiratory Illness Treatment (DART) program. The DART QI program is a multifaceted, web-based intervention that is delivered asynchronously over a 9-month period and takes a total of 2 hours to complete. DART's content is based on over a decade of observational research conducted by Mangione-Smith et al focused on optimizing provider-parent communication during pediatric ARTI visits in order to reduce unnecessary antibiotic prescribing while still maintaining parent satisfaction with care.[cites] The DART program also includes content related to evidence-based antibiotic prescribing with a particular focus on reducing the use of second-line, broad-spectrum antibiotics for bacterial ARTIs.

Under funding from the Eunice Kennedy National Institute for Child Health and Human Development (NICHD), the investigators recently conducted a trial of the DART QI program with 55 providers from 20 practices belonging to one of two pediatric practice-based research networks: the Pediatric Research in Office Settings (PROS) and NorthShore University Health System networks. Exposure to the DART QI program resulted in an proportional decrease from for overall antibiotic prescribing rates for ARTIs and a proportional decrease from for the use of second-line antibiotics for bacterial ARTIs comparing the baseline to the post-intervention periods.

The DART QI Program represents a new, innovative tool to address antibiotic over-use for ARTIs in the pediatric outpatient setting. However, it is unclear whether the program will be effective when disseminated to the family practice clinical setting where 23% of children receive their acute illness care nationally. It is also unclear how exposure to the communication strategies outlined in the DART QI program may influence provider-patient communication during adult encounters for ARTI.

ELIGIBILITY:
Inclusion Criteria:

1. Children or adults with acute respiratory tract infections (ARTIs) defined as bacterial (acute otitis media [AOM], pharyngitis, and sinusitis) or viral (bronchitis and viral upper respiratory infection [URI]) based on their common etiologies.
2. Seven months old and older

Exclusion Criteria:

1. 0 - 6 months old

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Overall antibiotic prescribing rates for pediatric and adult ARTIs. | The primary outcomewill be collected for all participating providers (both intervention and control) during a 30-month period beginning with baseline data collection.
  The primary outcome of overall antibiotic prescribing rates for ARTIs will be assessed by calculating the number of eligible ARTI visits occurring within a measurement period (measure denominator) where antibiotics were prescribed (numerator). This outcome will be assessed separately for the eligible pediatric (6 months to 17 years-old) and adult (> 18 years-old) patients.

SECONDARY OUTCOMES:
First-line antibiotic prescribing rates for pediatric and adult bacterial ARTIs. | The secondary outcome will be collected for all participating providers (both intervention and control) during a 30-month period beginning with baseline data collection.
  The secondary outcome of first-line antibiotic prescribing rates for bacterial ARTIs will be assessed by calculating the number of eligible bacterial ARTI visits occurring within a measurement period (measure denominator) where first-line antibiotics were prescribed (numerator). This outcome will be assessed separately for the eligible pediatric (6 months to 17 years-old) and adult (> 18 years-old) patients.
Net cost of delivering the DART QI program | This outcome will be collected for all participating providers (both intervention and control) during a 30-month period beginning with baseline data collection.
  The net cost of delivering the intervention will be calculated as the difference between the total costs (sum of antibiotic prescription, intervention delivery, and return visit utilization costs) in the intervention and control groups.

CONTACTS AND LOCATIONS:
Overall Officials: Rita Mangione-Smith, MD, MPH, Principal Investigator — Seattle Children's Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grijalva CG, Nuorti JP, Griffin MR. Antibiotic prescription rates for acute respiratory tract infections in US ambulatory settings. JAMA. 2009 Aug 19;302(7):758-66. doi: 10.1001/jama.2009.1163. PMID 19690308
- [Background] Hersh AL, Shapiro DJ, Pavia AT, Shah SS. Antibiotic prescribing in ambulatory pediatrics in the United States. Pediatrics. 2011 Dec;128(6):1053-61. doi: 10.1542/peds.2011-1337. Epub 2011 Nov 7. PMID 22065263
- [Background] Kronman MP, Zhou C, Mangione-Smith R. Bacterial prevalence and antimicrobial prescribing trends for acute respiratory tract infections. Pediatrics. 2014 Oct;134(4):e956-65. doi: 10.1542/peds.2014-0605. Epub 2014 Sep 15. PMID 25225144
- [Background] Fleming-Dutra KE, Hersh AL, Shapiro DJ, Bartoces M, Enns EA, File TM Jr, Finkelstein JA, Gerber JS, Hyun DY, Linder JA, Lynfield R, Margolis DJ, May LS, Merenstein D, Metlay JP, Newland JG, Piccirillo JF, Roberts RM, Sanchez GV, Suda KJ, Thomas A, Woo TM, Zetts RM, Hicks LA. Prevalence of Inappropriate Antibiotic Prescriptions Among US Ambulatory Care Visits, 2010-2011. JAMA. 2016 May 3;315(17):1864-73. doi: 10.1001/jama.2016.4151. PMID 27139059
- [Background] Chung A, Perera R, Brueggemann AB, Elamin AE, Harnden A, Mayon-White R, Smith S, Crook DW, Mant D. Effect of antibiotic prescribing on antibiotic resistance in individual children in primary care: prospective cohort study. BMJ. 2007 Sep 1;335(7617):429. doi: 10.1136/bmj.39274.647465.BE. Epub 2007 Jul 26. PMID 17656505
- [Background] Costelloe C, Metcalfe C, Lovering A, Mant D, Hay AD. Effect of antibiotic prescribing in primary care on antimicrobial resistance in individual patients: systematic review and meta-analysis. BMJ. 2010 May 18;340:c2096. doi: 10.1136/bmj.c2096. PMID 20483949
- [Background] Goossens H, Ferech M, Vander Stichele R, Elseviers M; ESAC Project Group. Outpatient antibiotic use in Europe and association with resistance: a cross-national database study. Lancet. 2005 Feb 12-18;365(9459):579-87. doi: 10.1016/S0140-6736(05)17907-0. PMID 15708101
- [Background] Michaelidis CI, Fine MJ, Lin CJ, Linder JA, Nowalk MP, Shields RK, Zimmerman RK, Smith KJ. The hidden societal cost of antibiotic resistance per antibiotic prescribed in the United States: an exploratory analysis. BMC Infect Dis. 2016 Nov 8;16(1):655. doi: 10.1186/s12879-016-1990-4. PMID 27825306
- [Background] Centers for Disaese Control and Prevention Antibiotic resistance threats in the United States, 2013. 2013; http://www.cdc.gov/drugresistance/threat Accessed July 25, 2018.
- [Background] Vaz LE, Kleinman KP, Raebel MA, Nordin JD, Lakoma MD, Dutta-Linn MM, Finkelstein JA. Recent trends in outpatient antibiotic use in children. Pediatrics. 2014 Mar;133(3):375-85. doi: 10.1542/peds.2013-2903. Epub 2014 Feb 2. PMID 24488744
- [Background] Shapiro DJ, Hicks LA, Pavia AT, Hersh AL. Antibiotic prescribing for adults in ambulatory care in the USA, 2007-09. J Antimicrob Chemother. 2014 Jan;69(1):234-40. doi: 10.1093/jac/dkt301. Epub 2013 Jul 25. PMID 23887867
- [Background] Mangione-Smith R, McGlynn EA, Elliott MN, McDonald L, Franz CE, Kravitz RL. Parent expectations for antibiotics, physician-parent communication, and satisfaction. Arch Pediatr Adolesc Med. 2001 Jul;155(7):800-6. doi: 10.1001/archpedi.155.7.800. PMID 11434847
- [Background] Mangione-Smith R, Elliott MN, Stivers T, McDonald LL, Heritage J. Ruling out the need for antibiotics: are we sending the right message? Arch Pediatr Adolesc Med. 2006 Sep;160(9):945-52. doi: 10.1001/archpedi.160.9.945. PMID 16953018
- [Background] Mangione-Smith R, Zhou C, Robinson JD, Taylor JA, Elliott MN, Heritage J. Communication practices and antibiotic use for acute respiratory tract infections in children. Ann Fam Med. 2015 May-Jun;13(3):221-7. doi: 10.1370/afm.1785. PMID 25964399
- [Background] Gerber JS, Prasad PA, Fiks AG, Localio AR, Grundmeier RW, Bell LM, Wasserman RC, Keren R, Zaoutis TE. Effect of an outpatient antimicrobial stewardship intervention on broad-spectrum antibiotic prescribing by primary care pediatricians: a randomized trial. JAMA. 2013 Jun 12;309(22):2345-52. doi: 10.1001/jama.2013.6287. PMID 23757082
- [Background] Merriam SB, Cafrrarella RS. Learing in Adulthood. San Francisco, CA: Jossey-Bass; 2008.
- [Background] Davis DA, Thomson MA, Oxman AD, Haynes RB. Changing physician performance. A systematic review of the effect of continuing medical education strategies. JAMA. 1995 Sep 6;274(9):700-5. doi: 10.1001/jama.274.9.700. PMID 7650822
- [Background] Little P, Stuart B, Francis N, Douglas E, Tonkin-Crine S, Anthierens S, Cals JW, Melbye H, Santer M, Moore M, Coenen S, Butler C, Hood K, Kelly M, Godycki-Cwirko M, Mierzecki A, Torres A, Llor C, Davies M, Mullee M, O'Reilly G, van der Velden A, Geraghty AW, Goossens H, Verheij T, Yardley L; GRACE consortium. Effects of internet-based training on antibiotic prescribing rates for acute respiratory-tract infections: a multinational, cluster, randomised, factorial, controlled trial. Lancet. 2013 Oct 5;382(9899):1175-82. doi: 10.1016/S0140-6736(13)60994-0. Epub 2013 Jul 31. PMID 23915885
- [Background] Butler CC, Simpson SA, Dunstan F, Rollnick S, Cohen D, Gillespie D, Evans MR, Alam MF, Bekkers MJ, Evans J, Moore L, Howe R, Hayes J, Hare M, Hood K. Effectiveness of multifaceted educational programme to reduce antibiotic dispensing in primary care: practice based randomised controlled trial. BMJ. 2012 Feb 2;344:d8173. doi: 10.1136/bmj.d8173. PMID 22302780
- [Background] Stivers T. Non-antibiotic treatment recommendations: delivery formats and implications for parent resistance. Soc Sci Med. 2005 Mar;60(5):949-64. doi: 10.1016/j.socscimed.2004.06.040. PMID 15589666
- [Background] Pace WD, Cifuentes M, Valuck RJ, Staton EW, Brandt EC, West DR. An electronic practice-based network for observational comparative effectiveness research. Ann Intern Med. 2009 Sep 1;151(5):338-40. doi: 10.7326/0003-4819-151-5-200909010-00140. Epub 2009 Jul 28. PMID 19638402
- [Background] Ajzen I, Madden TJ. Prediction of goal-directed behavior: attitudes, intentions, and perceived behavioral control. Journal lof Experimental Social Psychology. 1986;22:453-474.
- [Background] Simon TD, Cawthon ML, Stanford S, Popalisky J, Lyons D, Woodcox P, Hood M, Chen AY, Mangione-Smith R; Center of Excellence on Quality of Care Measures for Children with Complex Needs (COE4CCN) Medical Complexity Working Group. Pediatric medical complexity algorithm: a new method to stratify children by medical complexity. Pediatrics. 2014 Jun;133(6):e1647-54. doi: 10.1542/peds.2013-3875. Epub 2014 May 12. PMID 24819580
- [Background] Moher D, Hopewell S, Schulz KF, Montori V, Gotzsche PC, Devereaux PJ, Elbourne D, Egger M, Altman DG; Consolidated Standards of Reporting Trials Group. CONSORT 2010 Explanation and Elaboration: Updated guidelines for reporting parallel group randomised trials. J Clin Epidemiol. 2010 Aug;63(8):e1-37. doi: 10.1016/j.jclinepi.2010.03.004. Epub 2010 Mar 25. PMID 20346624
- [Background] Simon TD, Haaland W, Hawley K, Lambka K, Mangione-Smith R. Development and Validation of the Pediatric Medical Complexity Algorithm (PMCA) Version 3.0. Acad Pediatr. 2018 Jul;18(5):577-580. doi: 10.1016/j.acap.2018.02.010. Epub 2018 Feb 26. PMID 29496546
- [Background] Deyo RA, Cherkin DC, Ciol MA. Adapting a clinical comorbidity index for use with ICD-9-CM administrative databases. J Clin Epidemiol. 1992 Jun;45(6):613-9. doi: 10.1016/0895-4356(92)90133-8. PMID 1607900
- [Background] Quan H, Sundararajan V, Halfon P, Fong A, Burnand B, Luthi JC, Saunders LD, Beck CA, Feasby TE, Ghali WA. Coding algorithms for defining comorbidities in ICD-9-CM and ICD-10 administrative data. Med Care. 2005 Nov;43(11):1130-9. doi: 10.1097/01.mlr.0000182534.19832.83. PMID 16224307
- [Background] Gelman A, Hillman J. Data analysis using regression and multilevel/hierarchical models. Cambridge: Cambridge University Press; 2007.
- [Background] Goldstein H. Multilevel statistical models. 4th ed: Wiley; 2010.
- [Background] Raudenbush SW, Bryk AS. Heirarchical linear models: applications and data analysis methods. 2nd ed: Sage; 2002.
- [Background] Wright DR, Taveras EM, Gillman MW, Horan CM, Hohman KH, Gortmaker SL, Prosser LA. The cost of a primary care-based childhood obesity prevention intervention. BMC Health Serv Res. 2014 Jan 29;14:44. doi: 10.1186/1472-6963-14-44. PMID 24472122
- [Background] Xu X, Grossetta Nardini HK, Ruger JP. Micro-costing studies in the health and medical literature: protocol for a systematic review. Syst Rev. 2014 May 21;3:47. doi: 10.1186/2046-4053-3-47. PMID 24887208
- [Background] Drummond MF, Sculpher MJ, Torrance GW, O'Brien BJ, Stodart GL. Methods of economic evaluation of health care programmes. 3rd ed. New York: Oxford University Press; 2005.
- [Background] Jenkins TC, Irwin A, Coombs L, Dealleaume L, Ross SE, Rozwadowski J, Webster B, Dickinson LM, Sabel AL, Mackenzie TD, West DR, Price CS. Effects of clinical pathways for common outpatient infections on antibiotic prescribing. Am J Med. 2013 Apr;126(4):327-335.e12. doi: 10.1016/j.amjmed.2012.10.027. PMID 23507206
- [Background] Pihlajamaki M, Kotilainen P, Kaurila T, Klaukka T, Palva E, Huovinen P; Finnish Study Group for Antimicrobial Resistance (FiRe-Network). Macrolide-resistant Streptococcus pneumoniae and use of antimicrobial agents. Clin Infect Dis. 2001 Aug 15;33(4):483-8. doi: 10.1086/322735. Epub 2001 Jul 20. PMID 11462184
- [Background] Brennan-Krohn T, Ozonoff A, Sandora TJ. Adherence to guidelines for testing and treatment of children with pharyngitis: a retrospective study. BMC Pediatr. 2018 Feb 9;18(1):43. doi: 10.1186/s12887-018-0988-z. PMID 29426305
- [Background] Hersh AL, Shapiro DJ, Pavia AT, Fleming-Dutra KE, Hicks LA. Geographic Variability in Diagnosis and Antibiotic Prescribing for Acute Respiratory Tract Infections. Infect Dis Ther. 2018 Mar;7(1):171-174. doi: 10.1007/s40121-017-0181-y. Epub 2017 Dec 22. PMID 29273976
- [Background] Gerber JS, Prasad PA, Russell Localio A, Fiks AG, Grundmeier RW, Bell LM, Wasserman RC, Keren R, Zaoutis TE. Variation in Antibiotic Prescribing Across a Pediatric Primary Care Network. J Pediatric Infect Dis Soc. 2015 Dec;4(4):297-304. doi: 10.1093/jpids/piu086. Epub 2014 Oct 30. PMID 26582868
- [Background] Barnett ML, Linder JA. Antibiotic prescribing for adults with acute bronchitis in the United States, 1996-2010. JAMA. 2014 May 21;311(19):2020-2. doi: 10.1001/jama.2013.286141. No abstract available. PMID 24846041
- [Background] Hersh AL, Fleming-Dutra KE, Shapiro DJ, Hyun DY, Hicks LA; Outpatient Antibiotic Use Target-Setting Workgroup. Frequency of First-line Antibiotic Selection Among US Ambulatory Care Visits for Otitis Media, Sinusitis, and Pharyngitis. JAMA Intern Med. 2016 Dec 1;176(12):1870-1872. doi: 10.1001/jamainternmed.2016.6625. No abstract available. PMID 27775770
- [Background] Tyrstrup M, Melander E, Hedin K, Beckman A, Molstad S. Children with respiratory tract infections in Swedish primary care; prevalence of antibiotic resistance in common respiratory tract pathogens and relation to antibiotic consumption. BMC Infect Dis. 2017 Sep 4;17(1):603. doi: 10.1186/s12879-017-2703-3. PMID 28870173
- [Background] Cabral C, Horwood J, Hay AD, Lucas PJ. How communication affects prescription decisions in consultations for acute illness in children: a systematic review and meta-ethnography. BMC Fam Pract. 2014 Apr 8;15:63. doi: 10.1186/1471-2296-15-63. PMID 24708839
- [Background] Stivers T, Mangione-Smith R, Elliott MN, McDonald L, Heritage J. Why do physicians think parents expect antibiotics? What parents report vs what physicians believe. J Fam Pract. 2003 Feb;52(2):140-8. PMID 12585992
- [Background] Basu, A. Estimating costs and valuations of non-health benefits. 2nd ed. New York: Oxford University Press; 2017.
- [Background] Drummond MF, Sculpher MJ, Claxton K, Stoddart GL, Torrance GW. Methods for Economic Evaluation of Health Care Programmes. New York: Oxford University Press; 2015.
- [Background] Tang S. Profile of Pediatric Visits 2004-2007. American Academy of Pediatrics, 2010.
- See also: Mangione-Smith R. Dialogue Around Respiratory Treatment (DART). 2018; Accessed 07/31/18. — https://clinicaltrials.gov/ct2/show/study/NCT02943551?term=Mangione-Smith&rank=1
- See also: CAHPS 2.0 Questionnaires. 2007 — https://www.ahrq.gov/cahps/surveys-guidance/cg/visit/index.html
- See also: CMS Physician Fee Schedule. Accessed 9/14/18. — http://www.cms.gov/apps/physician-fee-schedule/overview.aspx